CLINICAL TRIAL: NCT06365827
Title: Investigation of Perioperative Assessed Biomarker I-FABP (Intestinal Fatty Acid-binding Protein) Level for Prediction of Acute Mesenteric Ischemia and Its Correlation With Acute Kidney Injury Followed by Extracorporeal Circulation
Brief Title: Perioperatively Assessed Biomarker I-FABP Level for Prediction of Acute Mesenteric Ischemia and Its Correlation With Acute Kidney Injury, Followed by Extracorporeal Circulation (aMIKI)
Acronym: aMIKI
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ293/20
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass; Acute Mesenteric Ischemia; Acute Kidney Injury; Non-Occlusive Mesenteric Ischaemia
Keywords: Extracorporeal circulation; intestinal fatty acid-binding protein; I-FABP; acute mesenteric ischemia; acute kidney injury; non-occlusive mesenteric ischemia (NOMI); Cystatin C; NGAL
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood (serum and citrate) aliquots Urine aliquots
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMI vs. non-AMI: AMI, those with a acute mesenteric ischemia vs. non-AMI, those without a condition
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — no intervention of interest

SUMMARY:
Acute mesenteric ischemia (AMI) is a severe condition that might occur after cardiovascular surgery. Several risk factors for AMI, such as multimorbidity, the use of vasopressors, and an increase in inflammatory markers have been identified in the past. However, these risk factors also seem to influence the blood and urine levels of I-FABP. This prospective pilot study intends to evaluate the value of perioperatively assessed I-FABP levels and to correlate these values with clinical or angiographic findings in mesenteric ischemia to improve a standardised diagnosis.

DETAILED DESCRIPTION:
Extracorporeal circulation (ECC) in the form of cardiopulmonary bypass (CPB) counts among the contemporary strategies for organ protection during major cardiovascular surgery. Despite protecting the organs from severe ischemia-reperfusion injury, it generates a significant inflammatory response that may produce organ dysfunction. An aortic cross-clamp is a key step in open cardiovascular surgery to interrupt the blood flow across the aorta for operation. After aortic cross-clamp release, peripheral vascular resistance decreases by 70 to 80%, causing hypotension in the lower half of the body. During the ischemia-reperfusion period Oxygen-free radicals and inflammatory cytokines produced, which may contribute to inflammation-induced tissue injury. As an inflammatory reaction after the cardiac surgery involving CPB, capillary leak syndrome is associated with increased morbidity and mortality. Microcirculatory alterations in the mesenteric artery during or after CPB contribute to the intestinal hypoperfusion. A suboptimal microperfusion and ischemia-reperfusion of the intestinal tissue during ECC are the trigger of altered gut permeability and a systemic inflammatory response syndrome in turn. The main mechanism of intestinal ischemia after Cardiovascular surgery is a non-occult mesenteric ischemia (NOMI). Contrarily to occlusive mesenteric ischemia by emboli or thrombosis, NOMI is related to a reduction in the splanchnic blood flow. NOMI is considered to be a rare (incidence around 1%) but severe and very often fatal complication after a cardiac surgery with a mortality rate up to 90%, in which the perfusion of the intestine is limited. In the diagnosis of a NOMI, an invasive angiography with a digital subtraction angiography (DSA) is considered to be the gold standard. And a common therapy for it is to correct the underlying vascular pathology and diffuse vasospasm with application of vasodilators. That is performed through an angiographically and precisely placed catheter in the superior mesenteric artery. clinical appearance of NOMI presents a myriad of symptoms and can be confusing, or might even be completely masked. In addition, there is still a lack of highly sensitive and specific biomarkers to predict the NOMI.

Furthermore, patients with postoperative NOMI had significantly high coincidence for acute kidney injury (AKI). NOMI has also been shown to correlate with renal insufficiency. Metzger et al. hypothesised that similar Pathophysiological mechanisms may trigger AKI in association with NOMI.

The aim of the study is to prospectively evaluate the level of perioperatively assessed I-FABP tests for NOMI and to correlate those with clinical or angiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing cardiac or vascular surgery with extracorporeal circulation

Exclusion Criteria:

* endocarditis or bacterial sepsis,
* hepatitis or HIV on the patient's medical history,
* cases in which informed consent to participate in the study could not be obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing cardiac or vascular surgery with extracorporeal circulation in University Hospital Giessen
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of I-FABP values with/and without acute mesenteric ischemia | 24 hours before and 36 hours after surgery
  Is the variation of I-FABP values different in patients with and without the mesenteric ischemia at the time of initial clinical suspicion?

SECONDARY OUTCOMES:
Time interval to mesenteric ischemia | 24 hours before until day 7 post-surgery
  How does the time interval between the incident of mesenteric ischemia and the measured I-FABP tests affect the result?
Overall mortality rate | until day 30 post-surgery
  Overall mortality rate until day 30
Correlation of I-FABP with biomarkers of acute kidney injury | 24 hours before until day 7 post-surgery
  How does the value of I-FABP correlate with acute kidney injury?
Association of mesenteric ischemia with hypercoagulable states | 24 hours before until day 7 post-surgery
  Can an increased I-FABP level in blood and urine be a predictor for procoagulatory state measured with thrombin generation assay?

OTHER OUTCOMES:
Incidence of stroke | until day 30 post-surgery
  incidence of stroke within 30 days post-surgery will be assessed
Association of I-FABP level and multi-organ failure or cardiovascular mortality | until day 30 post surgery
  Is an elevated I-FABP level associated with an increased risk for multiorgan failure or cardiovascular mortality?

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Giessen, Cardiovascular surgery, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided